CLINICAL TRIAL: NCT02669940
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C in the Russian Federation - An Observational, Multi-Center Study
Brief Title: Observational, Multi-Center Study of the Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C in the Russian Federation
Acronym: HCV RWE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-743
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-07

CONDITIONS: Chronic Hepatitis C; Genotype 1
Keywords: Ombitasvir; Dasabuvir; Paritaprevir
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With Chronic Hepatitis C Genotype 1: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir ± RBV according to standard of care and in line with the current local label.

SUMMARY:
This study seeks to assess the effectiveness, patient reported outcomes, work productivity and healthcare resource utilization of the interferon-free regimen of paritaprevir /ritonavir (r) - ombitasvir, ± dasabuvir ± ribavirin (RBV) in participants with chronic hepatitis C in a real life setting across clinical practice populations.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for observation in this cohort if the following applies:

* Treatment-naïve or -experienced adult male or female patients with confirmed chronic hepatitis C, genotype 1, receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir ± RBV according to standard of care and in line with the current local label
* If RBV is co-administered with paritaprevir/r - ombitasvir with or without dasabuvir, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)
* Patients must voluntarily sign and date informed consent prior to inclusion into the study

Exclusion Criteria:

* Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve or -experienced adult male or female patients with confirmed chronic hepatitis C genotype 1, receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir ± RBV according to standard of care and in line with the current local label.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovschikov, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/ritonavir [r] - ombitasvir with or without dasabuvir with ribavirin (RBV) according to standard of care and in line with the current local label.
- Paritaprevir/r - Ombitasvir, ± Dasabuvir - RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir without RBV according to standard of care and in line with the current local label.
Period: Overall Study
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir - RBV
Started | 63 | 95
Completed | 62 | 92
Not Completed | 1 | 3
Not completed — Failure to return | 0 | 3
Not completed — Insufficient follow-up data | 1 | 0

BASELINE CHARACTERISTICS:
Population: Core population: eligible, enrolled participants with known fibrosis status who started the treatment combination recommended in the current local label for their disease characteristics, and remained on treatment for > 55 days (for 12-week treatment) or > 139 days (for 24-week treatment).
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir with RBV according to standard of care and in line with the current local label.
- Total: Total of all reporting groups
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir - RBV | Total
Number analyzed (Participants) | 63 | 93 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.38) | 46.2 (11.59) | 48.1 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 45 | 79
  Male | 29 | 48 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 1 | 1 | 2
  White/Caucasian | 62 | 92 | 154

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-Treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) levels < 50 IU/mL 12 weeks after the last actual dose of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Core population: eligible, enrolled participants with known fibrosis status who started the treatment combination recommended in the current local label for their disease characteristics, and remained on treatment for >55 days (for 12-week treatment) or >139 days (for 24-week treatment). Subgroup: excludes participants with missing SVR12 results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir with or without RBV according to standard of care and in line with the current local label.
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 22.2 [12.7 to 34.5] | 16.1 [9.3 to 25.2] | 18.6 [12.8 to 25.6]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 23.3 [13.4 to 36.0] | 17.0 [9.9 to 26.6] | 19.6 [13.5 to 26.9]

2. Secondary Outcome: Percentage of Participants Meeting SVR12 Non-Response Categories of Breakthrough, Failure to Suppress, and/or Relapse
Description: Breakthrough is defined as at least 1 documented HCV RNA <50 IU/mL followed by HCV RNA ≥50 IU/mL during treatment. Failure to suppress is defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL. Relapse is defined as HCV RNA < 50 IU/mL at end of treatment or at the last on-treatment HCV RNA measurement followed by HCV RNA ≧ 50 IU/mL posttreatment.
Time Frame: 12 weeks after last actual dose of study drug
Population: Core population: eligible, enrolled participants with known fibrosis status who started the treatment combination recommended in the current local label for their disease characteristics, and remained on treatment for > 55 days (for 12-week treatment) or > 139 days (for 24-week treatment). Subgroup: excludes participants with missing SVR12 results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir with RBV according to standard of care and in line with the current local label.
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir without RBV according to standard of care and in line with the current local label.
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 73.0 [60.3 to 83.4] | 78.5 [68.8 to 86.3] | 76.3 [68.8 to 82.7]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 76.7 [64.0 to 86.6] | 83.0 [73.4 to 90.1] | 80.4 [73.1 to 86.5]

3. Secondary Outcome: SVR12 Non-Response: Percentage of Participants With Breakthrough
Description: Breakthrough is defined as at least 1 documented HCV RNA <50 IU/mL followed by HCV RNA ≥50 IU/mL during treatment.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 1.6 [0.0 to 8.5] | 3.2 [0.7 to 9.1] | 2.6 [0.7 to 6.4]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 1.7 [0.0 to 8.9] | 3.4 [0.7 to 9.6] | 2.7 [0.7 to 6.8]

4. Secondary Outcome: SVR12 Non-Response: Percentage of Participants With Failure to Suppress
Description: Failure to suppress is defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir) with RBV according to standard of care and in line with the current local label.
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir) with or without RBV according to standard of care and in line with the current local label.
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 61.9 [48.8 to 73.9] | 54.8 [44.2 to 65.2] | 57.7 [49.5 to 65.6]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 65.0 [51.6 to 76.9] | 58.0 [47.0 to 68.4] | 60.8 [52.5 to 68.7]

5. Secondary Outcome: SVR12 Non-Response: Percentage of Participants With Relapse
Description: Relapse is defined as HCV RNA <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA ≧ 50 IU/mL posttreatment.
Time Frame: 12 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 9.5 [3.6 to 19.6] | 20.4 [12.8 to 30.1] | 16.0 [10.6 to 22.7]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 10.0 [3.8 to 20.5] | 21.6 [13.5 to 31.6] | 16.9 [11.2 to 23.9]

6. Secondary Outcome: SVR12 Non-Response: Percentage of Participants With Premature Study Drug Discontinuation With No On-Treatment Virologic Failure
Description: On-treatment virologic failure included virological breakthrough and failure to suppress. Virological breakthrough was defined as at least one documented HCV RNA < 50 IU/mL or undetectable/negative followed by HCV RNA ≥ 50 IU/mL during treatment. Failure to suppress was defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL or positive.
Time Frame: 12 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV: Participants with confirmed chronic hepatitis C genotype 1 receiving combination therapy with paritaprevir/r - ombitasvir with or without dasabuvir) without RBV according to standard of care and in line with the current local label.
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 0 [0.0 to 5.7] | 0 [0.0 to 3.9] | 0 [0.0 to 2.3]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 0 [0.0 to 6.0] | 0 [0.0 to 4.1] | 0 [0.0 to 2.5]

7. Secondary Outcome: SVR12 Non-Response: Percentage of Participants With Missing SVR12 Data
Time Frame: 12 weeks after last actual dose of study drug
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants | 4.8 [1.0 to 13.3] | 5.4 [1.8 to 12.1] | 5.1 [2.2 to 9.9]

8. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks Post-Treatment (SVR24)
Description: SVR24 is defined as HCV RNA levels < 50 IU/mL 24 weeks after the last actual dose of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV.
Time Frame: 24 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 20.6 [11.5 to 32.7] | 14.0 [7.7 to 22.7] | 16.7 [11.2 to 23.5]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 20.0 [10.8 to 32.3] | 13.6 [7.2 to 22.6] | 16.2 [10.7 to 23.2]

9. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response is defined as HCV RNA < 50 IU/mL.
Time Frame: From baseline until end of treatment (12 or 24 weeks after actual first dose)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 31.7 [20.6 to 44.7] | 30.1 [21.0 to 40.5] | 30.8 [23.6 to 38.6]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 31.7 [20.3 to 45.0] | 30.7 [21.3 to 41.4] | 31.1 [23.7 to 39.2]

10. Other Pre Specified Outcome: Percentage of Participants Achieving SVR12: Additional Analysis
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) levels < 50 IU/mL or undetectable/negative 12 weeks after the last actual dose of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 93.7 [84.5 to 98.2] | 93.5 [86.5 to 97.6] | 93.6 [88.5 to 96.9]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 98.3 [91.1 to 100] | 98.9 [93.8 to 100] | 98.6 [95.2 to 99.8]

11. Other Pre Specified Outcome: Percentage of Participants Meeting SVR12 Non-Response Categories of Breakthrough, Failure to Suppress, and/or Relapse: Additional Analysis
Description: Breakthrough is defined as at least 1 documented HCV RNA <50 IU/mL or undetectable/negative followed by HCV RNA ≥50 IU/mL or positive during treatment. Failure to suppress is defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL or positive. Relapse is defined as HCV RNA < 50 IU/mL or undetectable/negative at end of treatment or at the last on-treatment HCV RNA measurement followed by HCV RNA ≧ 50 IU/mL or positive posttreatment.
Time Frame: 12 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 1.6 [0.0 to 8.5] | 1.1 [0.0 to 5.8] | 1.3 [0.2 to 4.6]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 1.7 [0.0 to 8.9] | 1.1 [0.0 to 6.2] | 1.4 [0.2 to 4.8]

12. Other Pre Specified Outcome: SVR12 Non-Response: Percentage of Participants With Breakthrough: Additional Analysis
Description: Breakthrough is defined as at least 1 documented HCV RNA <50 IU/mL or undetectable/negative followed by HCV RNA ≥50 IU/mL or positive during treatment.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 0 [0.0 to 5.7] | 0 [0.0 to 3.9] | 0 [0.0 to 2.3]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 0 [0.0 to 6.0] | 0 [0.0 to 4.1] | 0 [0.0 to 2.5]

13. Other Pre Specified Outcome: SVR12 Non-Response: Percentage of Participants With Failure to Suppress: Additional Analysis
Description: Failure to suppress is defined as each measured on-treatment HCV RNA value ≥ 50 IU/mL or positive.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 1.6 [0.0 to 8.5] | 0 [0.0 to 3.9] | 0.6 [0.0 to 3.5]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 1.7 [0.0 to 8.9] | 0 [0.0 to 4.1] | 0.7 [0.0 to 3.7]

14. Other Pre Specified Outcome: SVR12 Non-Response: Percentage of Participants With Relapse: Additional Analysis
Description: Relapse is defined as HCV RNA < 50 IU/mL or undetectable/negative at end of treatment or at the last on-treatment HCV RNA measurement followed by HCV RNA ≧ 50 IU/mL or positive posttreatment.
Time Frame: 12 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 0 [0.0 to 5.7] | 1.1 [0.0 to 5.8] | 0.6 [0.0 to 3.5]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 0 [0.0 to 6.0] | 1.1 [0.0 to 6.2] | 0.7 [0.0 to 3.7]

15. Other Pre Specified Outcome: Percentage of Participants Achieving SVR24: Additional Analysis
Description: SVR24 is defined as HCV RNA levels < 50 IU/mL or undetectable/negative 24 weeks after the last actual dose of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV.
Time Frame: 24 weeks after last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 93.7 [84.5 to 98.2] | 92.5 [85.1 to 96.9] | 92.9 [87.7 to 96.4]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 95.0 [86.1 to 99.0] | 95.5 [88.8 to 98.7] | 95.3 [90.5 to 98.1]

16. Other Pre Specified Outcome: Percentage of Participants Achieving Virological Response at End of Treatment: Additional Analysis
Description: Virologic response is defined as HCV RNA < 50 IU/mL or undetectable/negative.
Time Frame: From baseline until end of treatment (12 or 24 weeks after actual first dose)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
Number analyzed (Participants) | 63 | 93 | 156
percentage of participants
  Core Population | 93.7 [84.5 to 98.2] | 95.7 [89.4 to 98.8] | 94.9 [90.1 to 97.8]
  Core Population Subgroup: number analyzed (Participants) | 60 | 88 | 148
  Core Population Subgroup | 95.0 [86.1 to 99.0] | 96.6 [90.4 to 99.3] | 95.9 [91.4 to 98.5]

ADVERSE EVENTS:
Time Frame: The observational period for participants receiving 12 weeks of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV was maximum 36 weeks (12 weeks treatment and 24 weeks posttreatment observation). For participants receiving 24 weeks of paritaprevir/r - ombitasvir, ± dasabuvir, ± RBV the observational period was maximum 48 weeks (24 weeks treatment and 24 weeks posttreatment observation).
Arm/Group | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/95 | 0/158
Serious Adverse Events (participants affected / at risk) | 2/63 | 0/93 | 2/156
Other Adverse Events (participants affected / at risk) | 14/63 | 16/95 | 30/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV (N=63) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV (N=93) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV (N=156)
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, + RBV (N=63) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, - RBV (N=95) | Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± RBV (N=158)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 7 | 6 | 13
Fatigue (General disorders) | 1 | 2 | 3
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 2 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT02669940/SAP_000.pdf
  • Study Protocol (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT02669940/Prot_001.pdf